CLINICAL TRIAL: NCT04877145
Title: Single Drill Vrs Sequential Drill Dental Implants Placement
Brief Title: Implant Placement Using a Newly Designed Single Drill Versus Conventional Sequential Drills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mortada, lecturer of periodontology and oral implantology - faculty of dentistry , Assiut University - Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17300587
Record Dates: First submitted 2021-05-01; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Implant Complication
Keywords: implants
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single drill (Experimental): one drill to place the implants 3.25mm diameter stainless steel drill was used.
  Interventions: Other: drill
- sequential drills (Active Comparator): For the control group, four drills (2.2mm, 2.75mm, 3.25mm and 4mm diameter),
  Interventions: Other: drill

INTERVENTIONS:
Other: drill — single 3.25 mm stainless steel drill

SUMMARY:
dental implants are usually placed by sequential set of drills which could increase the time of the surgery and could raise the temperature of the osteotomy preparation so a new drill was designed to place the implants fast and easy way

DETAILED DESCRIPTION:
Dental implant success is evident nowadays with the predictable functional and aesthetic results obtained . Simplified techniques and approaches are preferred for the convenience of both the patients and operators . Current research is focusing on decreasing the number of instruments used, shortening of the operation time and performing flapless approaches for implant placement whenever possible. This is done to reduce the postoperative complaints, such as pain, swelling and bleeding; thus decreasing the need for analgesics and minimising the occurrence of morbidity .

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria :

  * implant recipient sites free from any pathological conditions.
  * Patients who were cooperative, motivated and hygiene conscious were selected.
  * non smoker patients
* exclusion criteria :

  * Patients unable to undergo minor oral surgical procedures
  * patients with a history of drug abuse or catabolic drugs were not included.
  * Patients with a history of psychiatric disorder and those with unrealistic expectations about the aesthetic outcome of implant therapy were also excluded.
  * Patients with insufficient vertical inter-arch space, on centric occlusion, to accommodate the available restorative components .
  * Uncontrolled diabetic patients
  * Patient who had any systemic condition that may contraindicate implant therapy (impaired wound healing - bleeding disorders
  * patients who had any habits that might jeopardise the osseointegration process, such as heavy smoking and alcoholism.
  * Patients with para-functional habits that produce overload on the implant, such as bruxism and clenching were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
osseointegration of the dental implants | 6 months
  healing and union of the dental implants with the surrounding bone measured by torque wrench exceeds 30 N/CM

SECONDARY OUTCOMES:
mobility | 6 months
  the fixation of the implants checked by perio test M (-8- 0) INDICATES nonmobile
bone loss | 6 months , 1 ,2 and 3 years after function
  by periapical xray the bone loss measured from the platform of the implant if present unit of measurement : mm

CONTACTS AND LOCATIONS:
Overall Officials: amr ah zahran, phd, Study Director — professor of periodontology
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
after using the single drill compared with the sequential drill all the implants checked for osseointegration , mobility and bone loss after function

REFERENCES:
- [Background] La Du BN. The human serum paraoxonase/arylesterase polymorphism. Am J Hum Genet. 1988 Sep;43(3):227-9. No abstract available. PMID 2843045
- [Background] Bacci C, Lucchiari N, Frigo AC, Stecco C, Zanette G, Dotto V, Sivolella S. Temperatures generated during implant site preparation with conventional drilling versus single-drill method: an ex-vivo human mandible study. Minerva Stomatol. 2019 Dec;68(6):277-284. doi: 10.23736/S0026-4970.19.04142-6. PMID 32052615
- [Background] Abboud M, Delgado-Ruiz RA, Kucine A, Rugova S, Balanta J, Calvo-Guirado JL. Multistepped Drill Design for Single-Stage Implant Site Preparation: Experimental Study in Type 2 Bone. Clin Implant Dent Relat Res. 2015 Oct;17 Suppl 2:e472-85. doi: 10.1111/cid.12273. Epub 2014 Sep 29. PMID 25263993
- [Background] Lucchiari N, Frigo AC, Stellini E, Coppe M, Berengo M, Bacci C. In Vitro Assessment with the Infrared Thermometer of Temperature Differences Generated During Implant Site Preparation: The Traditional Technique Versus the Single-Drill Technique. Clin Implant Dent Relat Res. 2016 Feb;18(1):182-91. doi: 10.1111/cid.12246. Epub 2014 Jul 17. PMID 25040939